CLINICAL TRIAL: NCT04073381
Title: Application of Ergogenic Aids to the Prehabilitation of Abdominal Cancer Patients Undergoing Cancer Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Hirofumi Tanaka, Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-08-0110
Record Dates: First submitted 2019-07-08; First posted 2019-08-29 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Prehabilitation
Keywords: Blood Flow Restriction Training; Ergogenic Aids; Abdominal Cancer

STUDY DESIGN:
Intervention Model Description: 100 subjects between the ages of 18 and 90, who have GI cancer and will undergo surgery will be recruited for this study. 100 is an arbitrary number of participants. Due to this study design not being previously use before power analysis calculations were unable to made for key variables. All subjects will participate in the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabiliation Program (Experimental): 100 subjects between the ages of 18 and 90, who have GI cancer and will undergo surgery will be recruited for this study ad participate in the prescribed prehabilitation exercise and nutrition program.
  Interventions: Combination Product: Prehabilitation Program

INTERVENTIONS:
Combination Product: Prehabilitation Program — This is a 4 week prehabilitation program which uses both exercise and nutrition. Exercise will be prescribed at least 6 days a week. Three days a week , for 45 mins, participants will be asked to perform body, leg and arm exercises against light resistance while wearing pneumatic blood flow restriction arm and leg bands. minutes. On the alternate days participants will walk approximately 15 minutes while wearing the leg bands that restrict blood flow. Additionally, a nutrition supplement cocktail will be provided and should be taken every day within 1 hour after completing each exercise session. The 4 Week Nutrition (Sports Drink) Supplement Cocktail: will include whey protein (25 g/day), creatine monohydrate (8 g/day), and L-citrulline (5 g/day). The supplement mixture will be provided in daily packages by the investigators (nutrition supplements are not regulated by the FDA)

SUMMARY:
The purpose of the proposed study is to measure surgical recovery, including the length of hospital stay, incidence of perioperative complications, and mortality at 90 days post-surgery, in surgical patients with abdominal cancer. The investigators hypothesize that this prehabilitation program will improve recovery and reduce perioperative complications via the proposed prehabilitation intervention.

DETAILED DESCRIPTION:
The investigators propose that steps to augment and optimize the effectiveness of prehabilitation interventions for abdominal cancer patients may be found in the field of sport science. The investigators have identified two primary strategies to improve and optimize prehabilitation in patients with abdominal cancer: exercise and nutritional supplementation. A home-based exercise program incorporating both walking and resistance training will be performed with blood flow restriction training (BFR). BFR is a cutting-edge training modality that works by restricting blood flow out of the veins by using compression devices similar to traditional blood pressure cuffs (1). This training modality is frequently used by injured athletes for enhanced recovery (2). Muscle hypertrophy and increased muscle strength are more robust and achievable with BFR, even if exercises are performed at low to moderate intensities (2). Additionally, the implementation of a sports nutrition supplement cocktail, which will be provided simultaneously with the 4-week BFR exercise intervention, was developed to augment the effects of resistance exercise by increasing overall anabolism (3) and to remedy the catabolic state that cancer patients often experience (4). The nutrition supplement cocktail will include whey protein, creatine monohydrate, and L-citrulline.

ELIGIBILITY:
Inclusion Criteria:

* Patients certified by a surgeon to participate in this study;
* Patients between the ages of 18 and 90;
* Patients with GI cancer.

Exclusion Criteria: Patients with

* Uncontrolled or active angina;
* New York Heart Association Class 3 or 4 heart failure;
* A myocardial infarction within the last 6 months;
* Severe/ uncontrolled hypertension (systolic pressure ≥180 mmHg or diastolic pressure ≥120mmHg);
* Uncontrolled diabetes (fasting blood glucose >400 mg/dL);
* American Society of Anesthesiologists (ASA) health status grade IV-V.
* Severe orthopedic conditions that prohibit or impede exercise;
* Wheelchair dependence;
* Co-morbid medical conditions interfering with the ability to perform exercise; -Severely impaired ambulation (i.e. patients with uncontrolled neuromuscular disorders);
* History of Acute Deep Venous Thrombosis within the last 6 months;
* Inability to comply with exercise instructions upon evaluation; or
* Inability to provide an informed consent (dementia);
* Taking medication/supplements containing nitrites/nitrates;
* With allergies to creatine monohydrate;
* With allergies or intolerance to artificial sweeteners such as Sucralose, Xylitol, Aspartame, or Stevia;
* Simultaneous participation in a pharmacotherapy trial;
* Estimated glomerular filtration rate (EGFR) < 30 and not currently on dialysis.
* Pregnant or lactating women
* Dementia
* Mini Mental State Examination score of Severe Impairment (≤17), or
* Patients with severe depression.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Hospital Measures- Length of hospital stay | Through study completion, an average 1year
  Length of hospital stay
Hospital Measures- Emergency room visits | Through study completion, an average 1 year
  emergency room visits
Hospital Measures- Readmission | Through study completion, an average 1 year
  Readmission
Hospital Measures | Through study completion, an average 1 year
  Mortality

SECONDARY OUTCOMES:
Physical Fitness- Hand Grip | Baseline, 4 weeks, and 8 weeks
  Hand grip dynamometry
Physical Fitness- 6MWT | Baseline and 4 weeks
  6 minute walk test
Physical Fitness- TUG | Baseline, 4 weeks, and 8 weeks
  Timed up and go
Physical Fitness- SPPB | Baseline and 4 weeks
  Short Physical Performance Battery Assessing Lower Extremity Function
Body Composition | Baseline and 4 weeks
  DXA (dual energy X-ray absorptiometry) will be used to assess body composition.
Blood Work- AA | Baseline and 4 weeks
  Amino Acids
Blood Work- CRP | Baseline and 4 weeks
  C-Reactive protein (CRP)
Blood Work- IL6 | Baseline and 4 weeks
  Interleukin 6 (IL-6)
Blood Work- TNFalpha | Baseline and 4 weeks
  TNF-alpha
Questionnaires- Health Status | Baseline
  Health research questionnaire; self reported medical and health history of participant.
Questionnaires- IPAQ | Baseline and 8 weeks
  International Physical Activity Questionnaire; self reported time, frequency and duration of physical activity within the last 7 days.
Questionnaires- SF36 | Baseline, 4 weeks, and 8 weeks
  SF-36 Quality of Life. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Questionnaires- MMSE | Baseline
  Mini Mental State Examination (MMSE) 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Score is reported as 0-30 . 24-30 indicates no cognitive impairment, 18-23 indicates mild cognitive impairment, and 0-17 indicates severe cognitive impairment.
Questionnaires- FESI | Baseline, 4 weeks, and 8 weeks
  Falls Efficacy Scale-International; items are summed to calculate a range of total score from minimum 16 to maximum 64. The higher the score the greater the fear of falling.
Questionnaires- Nutrition | Baseline
  Dietary Food and Supplement Intake; self reported nutrition intake from 2 weekdays and one weekend.
Questionnaires- Charlson Comorbidity | Baseline
  Charlson Comorbidity Index predicts the one-year mortality for a patient who may have a range of comorbid conditions, such as heart disease, AIDS, or cancer (a total of 22 conditions). Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. Scores are summed to provide a total score to predict mortality.
Questionnaires- BSCI | Baseline
  Brief Screen for Cognitive Impairment (BSCI); Scores are weighted and summed to arrive at final score. Delayed recall and medication help each get a weight of 2.0, and errand help gets a weight of 1.0. If client does not take any medications, the weighted scores of the other two items perform similarly to the three-item version. Higher scores indicate greater frailty/cognitive impairment.
Questionnaires- Edmonton Frailty | Baseline
  Edmonton Frailty Assessment; consists of nine domains and eleven items, each scoring 0 points (frailty absent or normal health), 1 point (minor errors or mild/moderate impairment), or 2 points (important errors or severely impaired). Higher scores indicate greater frailty.
Questionnaires- ECOG | Baseline
  Eastern Cooperative Oncology Group Performance Status; Determines ability of patient to tolerate therapies in serious illness, specifically for chemotherapy.
Questionnaires- Clock Test | Baseline
  Clock Test; evaluates three items: "correctly drawn clock shape," "all numbers in the correct position," and "hands of the clock set to the correct time." A score of 1 was assigned for each of these items. Higher scores indicate greater frailty/cognitive impairment.
Accerlometry | Through study completion, an average of one year
  Accelerometer/ Pedometer Measurement will be used to measure activity levels for 7 days immediately post surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Aging Research Laboratory at UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be reported as average group means.

REFERENCES:
- [Derived] Wooten SV, Wolf JS Jr, Mendoza D, Bartholomew JB, Stanforth PR, Stanforth D, Tanaka H, Fleming RYD. The Impact of a Multimodal Sport Science-Based Prehabilitation Program on Clinical Outcomes in Abdominal Cancer Patients: A Cohort Study. Am Surg. 2022 Sep;88(9):2302-2308. doi: 10.1177/00031348221103657. Epub 2022 May 24. PMID 35608376

DOCUMENTS (1):
  • Informed Consent Form (2020-05-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT04073381/ICF_000.pdf